CLINICAL TRIAL: NCT06285396
Title: Effect of Ephedrine, Phenylepinephrine, and Norepinephrine on Myometrial Contractility in Pregnant People With Type II and Gestational Diabetes During Cesarean Section: An In-vitro Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This was a undergraduate student project, with some preliminary results. It may or may not be continued in the future.
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-01
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Hemorrhage
Keywords: oxytocin; type II diabetes; gestational diabetes; uterine contraction
MeSH Terms: conditions — Postpartum Hemorrhage; Diabetes Mellitus, Type 2; Diabetes, Gestational | interventions — Ephedrine; Phenylephrine; Norepinephrine; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Control (No Intervention): The myometrial samples are bathed in physiological salt solution (PSS) only.
- Ephedrine (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of ephedrine.
  Interventions: Drug: Ephedrine
- Phenylephrine (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of phenylephrine.
  Interventions: Drug: Phenylephrine
- Norepinephrine (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of norepinephrine.
  Interventions: Drug: Norepinephrine
- Control + oxytocin (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) and oxytocin.
  Interventions: Drug: Oxytocin
- Ephedrine + oxytocin (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of ephedrine and oxytocin..
  Interventions: Drug: Ephedrine; Drug: Oxytocin
- Phenylephrine + oxytocin (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of phenylephrine and oxytocin..
  Interventions: Drug: Phenylephrine; Drug: Oxytocin
- Norepinephrine + oxytocin (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of norepinephrine and oxytocin..
  Interventions: Drug: Norepinephrine; Drug: Oxytocin

INTERVENTIONS:
Drug: Ephedrine — Ephedrine in solution, at applicable concentrations based on literature.
  Arms: Ephedrine; Ephedrine + oxytocin
Drug: Phenylephrine — Phenylephrine, at applicable concentrations based on literature.
  Arms: Phenylephrine; Phenylephrine + oxytocin
Drug: Norepinephrine — Norepinephrine, at applicable concentrations based on literature.
  Arms: Norepinephrine; Norepinephrine + oxytocin
Drug: Oxytocin — Oxytocin, at applicable concentrations based on literature.
  Other Names: pitocin
  Arms: Control + oxytocin; Ephedrine + oxytocin; Norepinephrine + oxytocin; Phenylephrine + oxytocin

SUMMARY:
The goal of this study is to learn about how medication that is used to help treat low blood pressure during a Cesarean delivery (CD) can cause changes to the uterine muscle tissue and its ability to contract, in patients with Type II and gestational diabetes.

Spinal anesthesia administered during elective CD has been known to cause hypotension (low blood pressure) as a side effect during the procedure, and is prevented by administration of vasopressors (medication to raise blood pressure) by the anesthesiologist after the delivery of the baby. Vasopressors treat hypotension by interacting with receptors on blood vessels that increase blood pressure, which can also cause changes to uterine contractility. Inadequate uterine contraction after CD can expose mothers to postpartum hemorrhage (PPH), with diabetic patients displaying a 2.5-times higher risk of PPH.

It is important to understand how vasopressor(s) might affect the uterine contractility of women with Type II and gestational diabetes. Since medication to contract the uterus is also routinely administered at delivery, it is important to study the effect of these drugs in combination. The purpose of this study is to compare uterine contractility patterns and receptor distribution in women with type II and gestational diabetic and control term pregnant patients with administration of vasopressors. This will be done using small uterine tissue samples taken from the incision site following CD, which will then be used for experiments in the laboratory.

DETAILED DESCRIPTION:
The global prevalence of diabetes has increased drastically over the past 20 years, with 1.5 million new cases each year. The prevalence of Type II diabetes in women of childbearing age has shown the greatest increase, in the United States alone rising from 33% in 1990-1998 to 70% in 2020. Additionally, the worldwide rate of cesarean delivery (CD) follows a similar trend. CD procedures can be both elective and emergent, with the rate of elective CD increasing by 30% in Canada since 2001. Neuraxial anesthesia administered during elective CD has been known to induce hypotension as a side effect, which is then countered by administering vasopressors such as epinephrine, norepinephrine, and phenylephrine that act on adrenergic alpha and beta receptors on smooth muscle tissue. However, since these receptors are expressed on the smooth muscle layer of the uterus called the myometrium, vasopressors can elicit changes in myometrial contractility. Inadequate myometrial contractility during CD can expose the mother to postpartum hemorrhage (PPH) which is a leading cause of maternal mortality worldwide.

Additionally, diabetic women undergoing CD are often obese (BMI > 30 kg/m2) or have macrosomia (larger than average baby), which are independent risk factors for PPH. However, there is still a 2.5-fold increased risk in PPH in Type II diabetic patients, even when adjusted for diabetic-associated obesity. Type II diabetics undergoing elective CD also display a reduced contractile profile (as previously explored through in-vitro calcium signaling), which may contribute to their increased risk of PPH. Current research on myometrial contractility shows that throughout the gestational period, the adrenergic receptor subtypes on the myometrial tissue may transition to more pro-contractile phenotypes, which may react differently to administered vasopressors and thus affect induced contractility during CD. Oxytocin, a uterotonic, is the standard treatment for preventing PPH administered immediately after delivery.

There is currently no literature on the unique effects of vasopressors to manage hypotension in obstetric patients who are diagnosed with Type II and gestational diabetes. The increased risk of PPH at CD seen in type II and Gestational diabetics mothers may be due to differences in adrenergic receptor distribution, which have different affinities to the vasopressors administered. No studies thus far have directly explored the role of vasopressors on myometrial contractions in this patient population.

As the use of a standardized vasopressor dosage becomes more routine during elective CD, it is important to understand how this will affect the myometrial contractility of women with Type II and gestational diabetes. The investigators hypothesize that administration of vasopressors in full term pregnant women with type II and gestational diabetes will cause decreased myometrial contractility compared to healthy controls, and that the diabetic tissue will possess a different adrenergic receptor subtype profile compared to controls.

Aim 1: Investigate the differences in myometrial contractility of type II and gestational diabetic vs. control term pregnant patients with administration of vasopressors

Aim 2: Determine the expression of adrenergic receptor subtypes on myometrium of term pregnant type II and gestational diabetic patients

Aim 3: Investigate the difference in downstream adrenergic pathways proteins in myometrial of type II and gestational diabetics vs control patients with administration of vasopressors

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given consent to participate in the study
* Patients with gestational age 37-41 weeks
* Patients previously diagnosed with either Type II or Gestational diabetes. For the healthy control group, no previous diagnosis is required for inclusion
* Patients of 19-45 years
* Patients of normal BMI (18-30 BMI) for the healthy control group only
* Baby is registered as normal weight for size for the healthy control group only
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring elective primary or first repeat caesarean delivery
* Patients undergoing caesarean delivery under spinal anesthesia

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients in labor and those receiving oxytocin for induction of labor
* Emergency caesarean delivery in labor
* Patients who have had previous uterine surgery involving myometrial dissection or >1 previous caesarean delivery
* Patients with risk factors for PPH such as those with polyhydramnios, preeclampsia, multiple gestation, morbid obesity, macrosomia (large for size baby), and previous history of PPH. However, for diabetic group, those with morbid obesity and macrosomia will not be excluded as these conditions are almost always associated with diabetes.
* For the healthy control group only, a BMI >30 or <18
* Maternal age >45

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Motility index | 4 hours
  Motility index (MI) is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  Frequency and amplitude are secondary outcome measures as described below.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 4 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 4 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist. The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No